CLINICAL TRIAL: NCT05238142
Title: In-Home Study With MiniMed™ 780G Pump Automated Control in Type 2 - Evaluation of the AHCL System in Adults With Insulin-requiring Type 2 Diabetes
Brief Title: In-Home Study With MiniMed™ 780G Pump Automated Control in Type 2-Evaluation of the AHCL System in Adults With Insulin-requiring Type 2 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Diabetes (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CIP341
Record Dates: First submitted 2022-02-03; First posted 2022-02-14 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2025-02

CONDITIONS: Type 2 Diabetes Treated With Insulin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- MiniMed 780G System (Experimental): Adult participants with insulin-requiring type 2 diabetes age 18-80 using the MiniMed 780G system for a combined run-in period and study period will be approximately 135 days long.
  Interventions: Device: MiniMed™ 780G Insulin Pump system

INTERVENTIONS:
Device: MiniMed™ 780G Insulin Pump system — MiniMed 780G insulin pump with Guardian 4 sensor (phase 1) MiniMed™ 780G BLE 2.0 insulin pump used in combination with Disposable Sensor 5 (phase 2)

SUMMARY:
The objective of the study is to assess the safety and effectiveness of MiniMed™ 780G system in adult subjects with insulin-requiring type 2 diabetes in a home setting. The combined run-in period and study period will be approximately 135 days long.

DETAILED DESCRIPTION:
Phase 1 of the study, will utilize the MiniMed™ 780G Insulin pump with Guardian 4 sensor for the run-in period, study period, and optional continued access. Phase 2 of the study will utilize the MiniMed™ 780G BLE2.0 insulin pump with the Disposable Sensor 5 for the run-in period and study period which will be approximately 135 days long. A total of up to 575 subjects with at least 300 subjects entering the study period of Phase 2, with insulin-requiring diabetes age 18-80 will be enrolled at up to 40 investigational centers across the United States.

ELIGIBILITY:
Inclusion Criteria:

1. Is age 18 - 80 years at time of screening.
2. Has a clinical diagnosis of type 2 diabetes for 2 years or more as determined via medical record or source documentation by an individual qualified to make a medical diagnosis.
3. Is on MDI regimen (basal/bolus regimen with long-acting insulin and rapid-acting analogs), defined as greater than or equal to 2 injections per day for at least 3 months prior signing the informed consent, or CSII pump therapy with or without CGM. The investigator will use their discretion to verify that insulin requirements have been stable for the last 3 months prior to screening.
4. Is able to comply with technology, according to Investigator's judgment
5. Does not require a legally authorized representative to consent on their behalf due to mental or intellectual disability.
6. Is willing to perform fingerstick blood glucose measurements as needed.
7. Is willing to wear the system continuously throughout the study.
8. Has a Glycosylated hemoglobin (HbA1c) of less than 10% (as processed by Central Lab) at time of screening visit.

   Note: All HbA1c blood specimens will be sent to and tested by a National Glycohemoglobin Standardization Program (NGSP) certified Central Laboratory. HbA1c testing must follow NGSP standards.
9. Has thyroid-stimulating hormone (TSH) in the normal range OR if the TSH is out of normal reference range the Free T3 is below or within the lab's reference range and Free T4 is within the normal reference range.
10. Is willing to upload data from the study pump, must have Internet access, and a computer system, or compatible smartphone that meets the requirements for uploading the study pump.
11. Is willing to take one of the following insulins and can financially support the use of insulin preparations as required by the study:

    1. Humalog (insulin lispro injection)
    2. NovoLog/NovoRapid (insulin aspart injection)
    3. Admelog (insulin lispro injection)

Exclusion Criteria:

1. Has a history of 2 or more episodes of severe hypoglycemia, which resulted in any the following during the 6 months prior to screening:

   1. Medical assistance (i.e., Paramedics, Emergency Room [ER] or Hospitalization)
   2. Coma
   3. Seizures
2. Has been hospitalized or has visited the ER in the 6 months prior to screening resulting in a primary diagnosis of uncontrolled diabetes.
3. Has had diabetic ketoacidosis (DKA) or hyperglycemic hyperosmolar syndrome (HHS) in the last 6 months prior to screening visit.
4. Will not tolerate tape adhesive in the area of sensor placement as assessed by a qualified individual.
5. Has any unresolved adverse skin condition in the area of sensor placement (e.g., psoriasis, dermatitis herpetiformis, rash, Staphylococcus infection) at time of screening.
6. Has (Total Daily Dose) of less than 8 units or greater than 250 units at time of screening.
7. Has positive GAD (Glutamic Acid Decarboxylase) Antibody test
8. Is female of child-bearing potential and result of pregnancy test is positive at screening
9. Is sexually active female of child-bearing potential and is not using a form of contraception deemed reliable by the investigator.
10. Is female and plans to become pregnant during the course of the study.
11. Is being treated for hyperthyroidism at time of screening.
12. Has diagnosis of adrenal insufficiency at time of screening.
13. Has taken any oral, injectable, or intravenous (IV) glucocorticoids within 8 weeks from time of screening visit, or plans to take any oral, injectable, or IV glucocorticoids during the course of the study.

    Note: Intra-articular injections to treat pain (e.g., joint pain, bursitis, etc.) are permitted
14. Is using hydroxyurea at time of screening or plans to use it during the study.
15. Is actively participating in an investigational study (drug or device) wherein he/she has received treatment from an investigational study drug or investigational study device in the last 2 weeks prior to screening.(Note: Did not apply to subjects who transitioned from Phase 1 to Phase 2)
16. Is currently abusing illicit drugs.
17. Is currently abusing marijuana.
18. Is currently abusing prescription drugs.
19. Is currently abusing alcohol.
20. Has a history of visual impairment which would not allow subject to participate in the study and perform all study procedures safely, as determined by the investigator.
21. Has elective surgery planned that requires general anesthesia during the course of the study.
22. Has sickle cell disease, hemoglobinopathy; or has received red blood cell transfusion or erythropoietin within 3 months prior to time of screening.
23. Plans to receive red blood cell transfusion or erythropoietin over the course of study participation.
24. Is diagnosed with current eating disorder such as anorexia or bulimia.
25. Has been diagnosed with chronic kidney disease greater than CKD2 that results in chronic anemia.
26. Has a hematocrit that is below the normal reference range of lab used.
27. Is on dialysis.
28. Has serum creatinine of >2 mg/dL.
29. Has celiac disease that is not adequately treated as determined by the investigator.
30. Has had any of the following cardiovascular events within 1 year of screening: myocardial infarction, unstable angina, coronary artery bypass surgery, coronary artery stenting, transient ischemic attack, cerebrovascular accident, angina, congestive heart failure, or ventricular rhythm disturbances.
31. Has had any of the following cardiovascular events 1 year or more prior to screening: Myocardial infarction, unstable angina, coronary artery bypass surgery, coronary artery stenting, transient ischemic attack, cerebrovascular accident, angina, congestive heart failure, or ventricular rhythm disturbances. Subject may be enrolled if clearance from a board-certified cardiologist is provided prior to or at Screening.
32. Is a member of the research staff involved with the study.
33. Has used a MiniMed 780G pump prior to screening (Note: In Phase 2, this applies to new subjects only).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 574 (Actual)
Dates: Start 2022-02-25 (Actual); Primary Completion 2025-01-11 (Actual); Study Completion 2025-01-11 (Actual)

PRIMARY OUTCOMES:
Primary Safety Endpoint - Change in HbA1c | 3 months
  The overall mean change in HbA1c from baseline to end of 3-month study period. Non-inferiority test.
Primary Effectiveness Endpoint - Percent of time in range (TIR 70-180 mg/dL) | 3 months
  The mean percent of time in range (TIR 70-180 mg/dL). Non-inferiority test.

SECONDARY OUTCOMES:
Secondary Effectiveness Endpoint - Percent of time in range (TIR 70-180 mg/dL) | 3 months
  The mean percent of time in range (TIR 70-180 mg/dL). Superiority test.

CONTACTS AND LOCATIONS:
Locations (31):
- United States (31):
  - Medical Investigations, Little Rock, Arkansas
  - Headlands Research California LLC, Escondido, California
  - Loma Linda University Medical Center, Loma Linda, California
  - Hoag Hospital Newport Beach, Newport Beach, California
  - Mills-Peninsula Medical Center: Diabetes Research Institute, San Mateo, California
  - Sansum Diabetes Research Institute, Santa Barbara, California
  - East Coast Institute for Research, Jacksonville, Florida
  - USF Diabetes Center, Tampa, Florida
  - Atlanta Diabetes Associates, Atlanta, Georgia
  - East Coast Institute for Research, Canton, Georgia
  - East Coast Institute for Research, Macon, Georgia
  - Endocrine Research Solutions, Roswell, Georgia
  - Javara, Thomasville, Georgia
  - NorthShore University Health System, Skokie, Illinois
  - Iowa Diabetes Research, West Des Moines, Iowa
  - MedStar Good Samaritan Hospital, Baltimore, Maryland
  - Endocrine & Metabolic Consultants, Rockville, Maryland
  - Park Nicollet International Diabetes Center, Saint Louis Park, Minnesota
  - Bryan Health, Lincoln, Nebraska
  - Atlantic Health System, Morristown, New Jersey
  - NYC Research Inc, Long Island City, New York
  - Northwell Health Physician Partners Endocrinology, New York, New York
  - Physicians East, Greenville, North Carolina
  - Texas Diabetes and Endocrinology, Austin, Texas
  - Javara, Conroe, Texas
  - Velocity Clinical Research, Dallas, Texas
  - Prime Revival Research Institute, Flower Mound, Texas
  - Houston Methodist Research Institute, Houston, Texas
  - Tekton Research, McKinney, Texas
  - Virginia Endocrinology Research, Chesapeake, Virginia
  - Rainier Clinical Research Center, Renton, Washington

IPD SHARING:
Plan to Share IPD: No